CLINICAL TRIAL: NCT05306041
Title: A Randomized, Open-label, Phase II Trial Comparing Neoadjuvant Endocrine Therapy in Combination with Trastuzumab, Pertuzumab +/- the PI3K Inhibitor Inavolisib in Patients with HER2-positive, HR-positive, PIK3CA Mutant Early Breast Cancer-GeparPiPPa
Brief Title: Neoadjuvant Endocrine Therapy +/- the PI3K Inhibitor Inavolisib in HER2+, HR+, PIK3CA Mutant Early Breast Cancer
Acronym: GeparPiPPa
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG105
Record Dates: First submitted 2022-03-09; First posted 2022-03-31 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: HER2-positive Breast Cancer
Keywords: GeparPiPPa; German Breast Group
MeSH Terms: interventions — inavolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inavolisib (Experimental): Inavolisib for 6 cycles (18 weeks) Neoadjuvant endocrine therapy in combination with dual anti-HER2 blockade consisting of ready-to-use fixed-dose combination of pertuzumab and trastuzumab as subcutaneous (PH-FDC SC) formulation q3w for 6 cycles (18 weeks)
  Interventions: Drug: Inavolisib; Drug: PHESGO; Drug: Endocrine therapy
- without Inavolisib (Other): Neoadjuvant endocrine therapy in combination with dual anti-HER2 blockade consisting of ready-to-use fixed-dose combination of pertuzumab and trastuzumab as subcutaneous (PH-FDC SC) formulation q3w for 6 cycles (18 weeks)
  Interventions: Drug: PHESGO; Drug: Endocrine therapy

INTERVENTIONS:
Drug: Inavolisib — daily application of 9 mg (may be decreased to 6 mg and to 3 mg)
  Arms: Inavolisib
Drug: PHESGO — fixed-dose combination of pertuzumab and trastuzumab with hyaluronidase s.c. (PH-FDC SC) q3w beginning on day 1 of cycle 1 for 6 cycles (18 weeks)
Drug: Endocrine therapy — Endocrine therapy per physician´s choice with either tamoxifen 20mg or an aromatase inhibitor +/- GnRH analogue for premenopausal women and men

SUMMARY:
Evaluation of the potential incremental efficacy and safety of inavolisib in the neoadjuvant endocrine treatment of early-stage HER2-positive, HR-positive, PIK3CA mutant breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, open-label, parallel-group, phase II study to evaluate the potential incremental efficacy and safety of inavolisib in the neoadjuvant treatment of early-stage HER2-positive, HR-positive, PIK3CA mutant breast cancer.

170 patients with confirmed eligibility criteria and PIK3CA mutant breast cancer will be randomized in a 1:1 ratio to receive: Neoadjuvant endocrine therapy in combination with dual anti-HER2 blockade consisting of ready-to-use fixed-dose combination of pertuzumab and trastuzumab as subcutaneous (PH-FDC SC) formulation q3w for 6 cycles (18 weeks) with (6cycles) or without inavolisib. Endocrine therapy consists of either tamoxifen 20mg or an aromatase inhibitor +/- GnRH analogue for premenopausal women and men.

In both study arms, treatment will be given until surgery/core-biopsy, disease progression, unacceptable toxicity, or withdrawal of consent of the patient.

All patients will undergo surgery or biopsy after completing study therapy to assess pCR rate.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent for all study procedures according to local regulatory requirements prior to beginning specific protocol procedures.
2. Untreated, unilateral primary carcinoma of the breast, confirmed histologically by core biopsy. Fine-needle aspiration alone is not sufficient. Incisional biopsy is not allowed.
3. Tumor lesion in the breast must be measurable in two dimensions, preferably by sonography.
4. Patients must be in the following stages of disease:

   • cT1b - cT3 regardless of nodal status In patients with multifocal or multicentric breast cancer the largest lesion (target lesion) should be measured.
5. HR+/HER2+ disease with centrally confirmed ER-status, PR-status, HER2-status, PIK3CA mutation (tumor), Ki-67 value and TILs on core biopsy (target lesion). ER/PgR positive and HER2-positive is defined according to current ASCO/CAP guidelines. Formalin-fixed, paraffin-embedded (FFPE) breast tissue from core biopsy of target lesion has therefore to be sent to the GBG central pathology laboratory prior to randomization. In patients with multifocal or multicentric breast cancer, all non-target lesions must also be HR+/HER2+, as confirmed by local testing.
6. Age ≥ 18 years, female and male.
7. ECOG Performance status 0-1.
8. Normal cardiac function must be confirmed by ECG and cardiac ultrasound (LVEF or shortening fraction) within 3 months prior to randomization. Results for LVEF must be above 55%.
9. Laboratory requirements:

   Hematology
   * Absolute neutrophil count (ANC) ≥ 1.5/ nL
   * Platelets ≥ 100/ nL and
   * Hemoglobin ≥ 10 g/dL (≥ 6.2 mmol/L) Hepatic function
   * Total bilirubin < ULN except for patients with Gilbert's syndrome who may only be included if the total bilirubin is ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN
   * AST and ALT ≤ 1.5x ULN and
   * Alkaline phosphatase ≤ 2.5x ULN

   Glucose Metabolism:

   • Glycosylated hemoglobin (HbA1c) < 6.5%
10. Negative pregnancy test (urine or serum) within 14 days prior to randomization for all women of childbearing potential. A woman is considered to be of childbearing potential if she is not hysterectomized or not postmenopausal.

    Postmenopausal is defined as:
    * ≥12 continuous months of amenorrhea with no identified cause other than menopause.
    * Having undergone bilateral oophorectomy.
11. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for least 7 months after the last dose of PH-FDC SC. Examples of non-hormonal contraceptive methods with a failure rate of < 1% per year include: bilateral tubal ligation; male partner sterilization; intrauterine devices. For men: men must remain abstinent or use a condom with a spermicidal product during the treatment period and for 7 months after the last dose of PH-FDC therapy to avoid exposing the embryo. Men and women must refrain from donating sperm/eggs during this same period.
12. Staging work-up according to country guidelines prior to randomization including:

    • Bilateral mammography and/or breast MRI in combination with a breast ultrasound. Exception: In men where MRI is medically not indicated breast ultrasound is sufficient.
13. Patient must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria

1. Patients with HER2-negative breast cancer and/or HER2-positive, HR-negative breast cancer.
2. Need of immediate neoadjuvant chemotherapy, e.g. inflammatory breast cancer.
3. Patients with definitive clinical or radiologic evidence of Stage IV cancer.
4. Excisional biopsy or lumpectomy and /or axillary lymph node dissection and/or sentinel lymph node biopsy performed prior to study entry (biopsy of clinical involved LN is warranted).
5. Prior chemotherapy or endocrine therapy or radiation therapy prior to study entry with the following exceptions:

   • If medically indicated, initiation of endocrine therapy up to 28 days prior to randomization and use of established fertility preservation methods in young patients interested in subsequent pregnancies is allowed.
6. Patients with a history of breast cancer are ineligible with the following exceptions:

   • Patient has been disease-free for more than 5 years and is at low risk for recurrence (at the investigator's discretion).
7. Patients with a history of any treated malignancy are ineligible in case of high risk of recurrence (at the investigator's discretion) and/or ongoing oncological treatment. This also applies to patients who are at high risk that oncological treatment is indicated during study therapy.
8. Patients with BMI>30 can be included at the investigator's discretion.
9. Known hypersensitivity reaction to one of the compounds or substances, and/or murine proteins, and/or recombinant human hyaluronidase used in this protocol.
10. Patients with an established diagnosis of diabetes mellitus type I or uncontrolled type II based on FPG and HbA1c.
11. Patients who are immunocompromised as the result of HIV or receiving immunosuppressive therapies.
12. Clinically significant and active liver disease, for example, sclerosing cholangitis, active viral hepatitis B or C infection, or autoimmune hepatic disorders.
13. Patients with inflammatory bowel disease, such as Crohn's disease or ulcerative colitis, and active bowel inflammation (e.g., diverticulitis).
14. Patients with any concurrent ocular or intraocular condition, excluding baseline cataracts, that would require medical or surgical intervention during the study period to prevent or treat vision loss. In addition, patients with active uveitis or vitritis, history of uveitis, or active infectious process in the eye.
15. Patients with currently documented pneumonitis/interstitial lung disease.
16. Known or suspected congestive heart failure (>NYHA I) and / or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, uncontrolled or poorly controlled arterial hypertension (i.e. BP >160 / 90 mm Hg under treatment with three antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease.
17. Damaged skin at planned site of subcutaneous (SC) injections (thigh).
18. Patients who may have had a recent episode of thromboembolism and are still trying to optimize the anticoagulation dose and/or have not normalized their INR.
19. Concurrent treatment with: • Chronic corticosteroids unless initiated > 6 months prior to study entry and at low dose (10 mg or less methylprednisolone or equivalent).

    * Sex hormones. Prior treatment must be stopped before randomization (GnRH a is allowed).
    * Other experimental drugs or any other anti-cancer therapy.
20. Participation in another clinical trial with any investigational, not marketed drug within 30 days prior to study entry.
21. Female patients: pregnancy or lactation at the time of randomization.
22. History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent.
23. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response in the breast and axillary lymph nodes (ypT0/is ypN0) | 21 weeks (time window + 3 weeks)
  Pathological complete response (ypT0/is ypN0) is defined as no microscopic evidence of residual invasive tumor cells in all resected specimens of the breast and axilla.

SECONDARY OUTCOMES:
Rates of ypT0 ypN0; ypT0 ypN0/+; ypT0/is ypN0/+; ypT(any) ypN0 | 21 weeks (time window + 3 weeks)
  ypT0 ypN0 is defined as no microscopic evidence of residual invasive or non-invasive viable tumor cells in all resected specimens of the breast and axilla; ypT0 ypN0/+ is defined as no microscopic evidence of residual invasive or non-invasive viable tumor cells in all resected specimens of the breast; ypT0/Tis ypN0/+ is defined as no microscopic evidence of residual invasive viable tumor cells in all resected specimens of the breast
pCR rates per arm separately for the stratified subpopulations | 21 weeks (time window + 3 weeks)
  Pathological complete response (ypT0/is ypN0) is defined as no microscopic evidence of residual invasive tumor cells in all resected specimens of the breast and axilla.
Response rates of the breast tumor and axillary nodes based on physical examination and imaging tests (sonography, mammography, or MRI) after study treatment in both arms | 21 weeks (time window + 3 weeks)
  Clinical (c) and imaging (i) response will be assessed every 2nd cycle and before surgery by physical examination and imaging tests. Sonography is the preferred examination.
  The response categories of the breast are:
  * Complete response (CR): complete disappearance of all tumor signs in the breast
  * Partial response (PR): reduction in the product of the two largest perpendicular diameters of the primary tumor size by 50% or more
  * Stable disease (NC): no significant change in tumor size during treatment which means an estimated reduction of the tumor area by less than 50%, or an estimated increase in the size of the tumor area lesions of less than 25%
  * Progressive disease (PD): development of new, previously undetected lesions, or an estimated increase in the size of pre-existing lesions by 25% or more after at least two cycles of therapy
Percentage of patients receiving additional neoadjuvant chemotherapy after residual disease was confirmed by core biopsy at the end of study treatment | 21 weeks (time window + 3 weeks)
  In case of ycT0 and no tumor residuals in the biopsy, it is recommended to undergo surgery. Further neoadjuvant or adjuvant treatment including chemotherapy, radiotherapy, endocrine therapy and HER2-therapy will be administered at the discretion of the investigator and according to standard of care.
Breast conservation rate after treatment | 21 weeks (time window + 3 weeks)
  Breast conservation is defined as tumorectomy, segmentectomy or quadrantectomy as a most radical surgery.
Safety and tolerability profile (haematological and non-haematological adverse events) after the first 20 and the first 40 patients who started therapy and have completed two cycles of therapy | 6 weeks
  Tolerability and safety analyses include assessment of patients whose treatment had to be dose reduced, delayed or permanently stopped. The reason for treatment discontinuation includes aspects of efficacy (e.g. discontinuation due to tumor progression), safety (e.g. discontinuation due to haematological and non-haematological adverse events) and compliance (e.g. discontinuation due to withdrawal of consent). Safety by toxicity grades are defined by the NCI-CTCAE version 5.0
Overall safety and tolerability and treatment compliance in the two arms | 21 weeks (time window + 3 weeks)
  Descriptive statistics for the 2 treatment arms will be given on the number of patients whose treatment had to be dose reduced, delayed or permanently stopped. Reasons for premature discontinuation will be categorized according to the main reason and will be presented in frequency tables. Safety by toxicity grades are defined by the NCI-CTCAE version 5.0, laboratory parameters will be converted in CTC-grades and reported together with other adverse events.
Invasive disease-free survival (IDFS) and overall survival (OS) in both arms and according to stratified subpopulations (data collected within a registry). | up to 5 years
  Survival endpoints are defined as the time period between randomization and first event and will be analyzed after the end of the study by referring to data from GBG´s registries

CONTACTS AND LOCATIONS:
Overall Officials: Mattea Reinisch, PD Dr. med., Principal Investigator — Universitätsmedizin Mannheim, Frauenklinik mit Brustzentrum
Locations (29):
- Germany (26):
  - KEM Kliniken Essen-Mitte, Essen, North Rhine-Westphalia
  - Hämatologie-Onkologie im Zentrum MVZ GmbH, Augsburg
  - DBZ Onkologie, Berlin
  - Praxisklinik Krebsheilkunde für Frauen, Berlin
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Department of Breast-Center Holweide - Kliniken der Stadt Köln, Cologne
  - Städtisches Klinikum Dessau, Dessau
  - University Hospital Carl Gustav Carus, Dresden
  - Center for Gynecologic Oncology, Düsseldorf
  - Frauenklinik des Universitätsklinikums Erlangen, Erlangen
  - Klinik für Gynäkologie und Geburtshilfe Agaplesion Markus Krankenhaus, Frankfurt
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Mammazentrum HH am Krankenhaus Jerusalem, Hamburg
  - Klinikum Hanau, Hanau
  - DIAKOVERE Henriettenstift Frauenklinik, Hanover
  - National Center for Tumor Diseases - University Hospital Heidelberg, Heidelberg
  - Elisabeth Krankenhaus Brustzentrum, Kassel
  - Praxis für Hämatologie und Onkologie Koblenz and InVo - Institut für Versorgungsforschung in der Onkologie GbR, Koblenz
  - University Hospital Mannheim, Mannheim
  - University Hospital Gießen and Marburg, Campus Marburg, Marburg
  - Media Vita GmbH (MVZ), Münster
  - University Hospital Tübingen, Tübingen
  - Department of Gynecology and Obstetrics - University of Ulm, Ulm
  - GRN Klinik Weinheim, Weinheim
  - Klinikum Worms, Worms
  - Helios Universitätsklinikum Wuppertal, Wuppertal
- Italy (3):
  - Università Politecnica delle Marche - Azienda Ospedaliero Universitarià delle Marche, Ancona
  - AULSS9 Scaligera - Ospedale Mater Salutis di Legnago, Legnago
  - Istituto Europeo di Oncologica, Milan

IPD SHARING:
Plan to Share IPD: No